CLINICAL TRIAL: NCT04824989
Title: Advancing Engagement and Efficacy of Interventions for Co-Morbid Sleep and Behavior Problems in Young Children
Brief Title: Parents Advancing Toddler Health
Acronym: PATH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston University Charles River Campus (Other)
Collaborators: University of Denver (Other); University of Michigan (Other); Denver Health and Hospital Authority (Other); University of Colorado, Boulder (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01HD098167-01A1 (NIH); 5554E (Other: Boston University)
Record Dates: First submitted 2021-03-10; First posted 2021-04-01 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Sleep Problem; Behavior, Child
Keywords: sleep problems; behavior problems; parenting interventions; early childhood; poverty
MeSH Terms: conditions — Parasomnias; Child Behavior; Mental Disorders | interventions — Oral Health

STUDY DESIGN:
Intervention Model Description: Families are randomly assigned to one of four groups for an 8-week parent coaching intervention program: focus on (1) child sleep, (2) child behavior, (3) parent choice of child sleep or child behavior, (4) active control - safety & hygiene
Who Masked: Outcomes Assessor
Masking Description: Assessors are blind to participant assignment. Participant and Care Provider cannot be blind as the assignment determines the focus of the intervention received (sleep, behavior, choice, or safety/hygiene).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sleep Health (Experimental): Family receives the Sleep Health In Preschoolers parenting intervention to address toddler sleep problems.
  Interventions: Behavioral: Sleep Health in Preschoolers (SHIP)
- Behavior Health (Experimental): Family receives the Family Check-Up parenting intervention to address toddler behavior problems.
  Interventions: Behavioral: Family Check-Up (FCU)
- Choice (Experimental): Family is given the opportunity to select either the Sleep Health in Preschoolers intervention to address toddler sleep problems or the Family Check-Up intervention to address toddler behavior problems.
  Interventions: Behavioral: Sleep Health in Preschoolers (SHIP); Behavioral: Family Check-Up (FCU)
- Control (Active Comparator): Family receives a safety and hygiene active control intervention.
  Interventions: Behavioral: Oral Health, Child Safety, and Environmental Health Intervention (Active Control)

INTERVENTIONS:
Behavioral: Sleep Health in Preschoolers (SHIP) — SHIP is an 8 session home visiting intervention to reduce child sleep problems using a framework that draws from motivational interviewing and social cognitive theory, and effectively improves sleep timing, duration, and quality. Following ecological assessment of child sleep and sleep routines, feedback is provided on family strengths and challenges in the child sleep domain, with motivational interviewing to increase parent knowledge of sleep, correct misperceptions, and raise outcomes expectations. The remaining sessions are targeted modules that give tailored feedback and education, and coach the parent in setting manageable goals, identifying action steps, anticipating barriers, and supporting positive behaviors. Targets: bedtime scheduling, consistency, and routines; media use, independent sleep onset, nightmares and fears, night wakings, and early waking; sleep location, nap issues, engaging other caregivers.
  Arms: Choice; Sleep Health
Behavioral: Family Check-Up (FCU) — FCU is an 8 session home visiting intervention to reduce behavior problems for children through improved parenting. Over 30 years of research establishes its efficacy in reducing behavioral and emotional problems, including in low income toddlers. Following ecological assessment of behavior management and child behavior, family receives feedback on family strengths and challenges within the behavioral domain via a motivational interviewing approach. The remaining sessions are targeted modules drawn from the Everyday Parenting curriculum, individualized based on parent goals and identified challenge areas. Each session begins by establishing a collaborative skill set, involves teaching the rationale for a skill, teaching and modeling effective use of the skill, and then role play and experiential practice to coach the parent to success. Targets can include Positive Behavior Support, Limit Setting and Monitoring, Family Routines, Communication, and Problem Solving.
  Arms: Behavior Health; Choice
Behavioral: Oral Health, Child Safety, and Environmental Health Intervention (Active Control) — This intervention serves as an active control condition to ensure that observed effects are due to the intervention content, rather than to study processes, staff attention, or general support and problem solving. The intervention is designed to be comparable to SHIP and FCU in intensity, personal contact, session structure and approach, but focused on Oral Health, Child Safety, and Environmental Health, domains which should not immediately affect study outcomes.
  Arms: Control

SUMMARY:
Although early interventions can improve health equity in young children living in poverty, this promise often is not realized because of barriers to family engagement. The proposed study will target co-morbid behavior and sleep problems in early childhood, comparing child outcomes and family response to sleep and behavior interventions and investigating the novel strategy of letting families select their intervention.We will enroll 500 low-income toddlers with co-morbid sleep and behavior problems, randomized to 4 parent coaching interventions: sleep, behavior, family choice (sleep or behavior), and an active control. At baseline and at 1, 5, and 9 months post- intervention, we will assess child sleep and behavior and family functioning. We will measure family preference, engagement, and perceived value of each intervention. The goals of the study are: (1) to examine effects of evidence- based sleep and behavior interventions in young low-income children with co-morbid sleep and behavior problems on child sleep and behavior and family functioning; (2) to determine whether parents prefer, engage with, and value a sleep or behavior intervention more; and (3) to examine if giving families a choice of intervention results in higher engagement, higher perceived value and better family and child outcomes than assignment to intervention. By informing best practices for engaging low-income families to treat co-morbid sleep and behavior problems, results will be critical to reducing health disparities for children living in poverty.

DETAILED DESCRIPTION:
Children living in poverty have a high incidence of early-developing sleep and behavior problems, which are often co-morbid. Early sleep and behavior problems are prevalent and persistent risk factors for lifelong poor mental and physical health outcomes, and may be key mechanisms underlying early and enduring socioeconomic health disparities. While effective interventions exist, low-income families have low enrollment and retention in these interventions. Stigma of treating behavior problems creates an additional barrier to treatment. This RCT aims to address these barriers to treatment for low-income children with co-morbid sleep and behavior problems. Sleep and behavior problems and family dysfunction transact across time, increasing in severity, while healthy sleep, positive child behaviors, and effective parenting can support each other across development. Thus we posit that intervention in one domain, either sleep or behavior, may improve outcomes both within and across domains.

The proposed study is a parallel randomized controlled trial of behavioral treatments for sleep problems and behavior problems in early childhood. The current study will test our three key aims: that evidence based sleep and behavior interventions each will improve trajectories from early comorbid sleep and behavior problems to healthier outcomes (Aim 1); that family preference, engagement, and value may differ for sleep vs. behavior interventions (Aim 2); and that families who choose between sleep and behavior interventions will have a more positive family response and better outcomes than those assigned to an intervention (Aim 3). This study will enroll 500 low income children ages 24 to 48 months with comorbid sleep and behavior problems. Children will be recruited at Boston University and the University of Denver. Eligible participants will be randomized to one of four intervention arms, Behavior (FCU), Sleep (SHIP), Choice (FCU or SHIP, as selected by primary caregiver), and active Control (Oral Health, Child Safety, and Environmental Health). For those assigned to Choice, the primary caregiver will be provided information about FCU and SHIP and will select their preferred intervention.

At the baseline evaluation (T1) all participants will undergo the following procedures: a) An evaluation of child behavior b) an evaluation of child sleep c) an evaluation of family functioning. Following the baseline evaluation all participants will engage in 8 sessions of parent coaching intervention over a 2 month period, with the content of the intervention varying by intervention arm, see descriptions below. The SHIP and FCU have similar structure, emphasizing motivational interviewing and support for parent goals. Paraprofessional staff at each site will be trained to deliver the FCU, SHIP, and Control interventions.

The measures included in the T1 baseline evaluation will be repeated at 1 and 5 months post intervention, T2 and T3. At T4, 9 months post intervention, primary caregiver report of child behavior and sleep symptoms and family functioning will be collected via telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* child age at enrollment of 18-48 months;
* household income at or below 300% of the federal poverty line
* a parent fluent in English or Spanish
* child behavior problem as indicated by a score > 60 on the Emotionally Reactive, Anxious/Depressed, Withdrawn, Attention Problems, or Aggressive Behavior subscales of the Child Behavior Checklist 1 ½ - 5 years (CBCL 1 ½ - 5)
* child sleep problem as indicated by at least one of the following: score 1 standard deviation above community means on any subscale of the Children's Sleep Wake Scale or on the Sleep Anxiety subscale of the Children's Sleep Habits Questionnaire; nighttime sleep latency longer than 30 minutes; score >40 on the Children's Sleep Habits Questionnaire (CSHQ); bedtimes or wake times varying by more than 2 hours from day to day; and/or nighttime sleep duration ≤ 9.5 hr.

Exclusion Criteria:

* Diagnosed developmental disabilities
* Serious chronic medical conditions such as autoimmune disorders or cancer
* A positive screen on the Sleep Disordered Breathing or Parasomnia subscales of the CSHQ or parent-reported diagnosis of obstructive sleep apnea

Ages: 18 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Child Behavior Checklist (CBCL) from screening to one month | Change from screening to one month post-intervention
  This parent report for ages 1.5-5 assesses clinically significant behavior problems and yields age-normed subscales
Change in Child Behavior Checklist (CBCL) from screening to five months | Change from screening to five months post-intervention
  This parent report for ages 1.5-5 assesses clinically significant behavior problems and yields age-normed subscales
Change in Child Behavior Checklist (CBCL) from screening to nine months | Change from screening to nine months post-intervention
  This parent report for ages 1.5-5 assesses clinically significant behavior problems and yields age-normed subscales
Change in Emotion Regulation Checklist (ERC) from baseline to one month | Change from baseline to one month post-intervention
  Parent report assessing intensity, flexibility, and appropriateness of child emotions
Change in Emotion Regulation Checklist (ERC) from baseline to five months | Change from baseline to five months post-intervention
  Parent report assessing intensity, flexibility, and appropriateness of child emotions
Change in Emotion Regulation Checklist (ERC) from baseline to nine months | Change from baseline to nine months post-intervention
  Parent report assessing intensity, flexibility, and appropriateness of child emotions
Change in Children's Sleep Wake Scale (CSWS) from screening to one month | Change from screening to one month post-intervention
  Parent report assessing child bedtime resistance, sleep quality, and daytime sleepiness
Change in Children's Sleep Wake Scale (CSWS) from screening to five months | Change from screening to five months post-intervention
  Parent report assessing child bedtime resistance, sleep quality, and daytime sleepiness
Change in Children's Sleep Wake Scale (CSWS) from screening to nine months | Change from screening to nine months post-intervention
  Parent report assessing child bedtime resistance, sleep quality, and daytime sleepiness
Change in nighttime sleep minutes from baseline to one month as measured by actigraphy | Change from baseline to one month post-intervention
  The Actiwatch Spectrum Plus actigraph will be worn on the child's non-dominant wrist for one week at each assessment to provide continuous recording of state via motion detection, and will yield an index of nighttime sleep minutes. Data are analyzed using Actiware software.
Change in nighttime sleep minutes from baseline to five months as measured by actigraphy | Change from baseline to five months post-intervention
  The Actiwatch Spectrum Plus actigraph will be worn on the child's non-dominant wrist for one week at each assessment to provide continuous recording of state via motion detection, and will yield an index of nighttime sleep minutes. Data are analyzed using Actiware software.
Change in sleep onset from baseline to one month as measured by actigraphy | Change from baseline to one month post-intervention
  The Actiwatch Spectrum Plus actigraph will be worn on the child's non-dominant wrist for one week at each assessment to provide continuous recording of state via motion detection, and will yield an index of sleep onset. Data are analyzed using Actiware software.
Change in sleep onset from baseline to five months as measured by actigraphy | Change from baseline to five months post-intervention
  The Actiwatch Spectrum Plus actigraph will be worn on the child's non-dominant wrist for one week at each assessment to provide continuous recording of state via motion detection, and will yield an index of sleep onset. Data are analyzed using Actiware software.
Change in sleep consistency from baseline to one month as measured by actigraphy | Change from baseline to one month post-intervention
  The Actiwatch Spectrum Plus actigraph will be worn on the child's non-dominant wrist for one week at each assessment to provide continuous recording of state via motion detection, and will yield an index of sleep consistency (consistency in sleep timing from night to night). Data are analyzed using Actiware software.
Change in sleep consistency from baseline to five months as measured by actigraphy | Change from baseline to five months post-intervention
  The Actiwatch Spectrum Plus actigraph will be worn on the child's non-dominant wrist for one week at each assessment to provide continuous recording of state via motion detection, and will yield an index of sleep consistency (consistency in sleep timing from night to night). Data are analyzed using Actiware software.

SECONDARY OUTCOMES:
Change in Children's Sleep Hygiene Scale (CSHS) from baseline to one month | Change from baseline to one month post-intervention
  Parent report assessing sleep inhibiting and sleep facilitating behaviors
Change in Children's Sleep Hygiene Scale (CSHS) from baseline to five months | Change from baseline to five months post-intervention
  Parent report assessing sleep inhibiting and sleep facilitating behaviors
Change in Children's Sleep Hygiene Scale (CSHS) from baseline to nine months | Change from baseline to nine months post-intervention
  Parent report assessing sleep inhibiting and sleep facilitating behaviors
Change in Parenting Sense of Competence (PSOC) from baseline to one month | Change from baseline to one month post-intervention
  Parent report assessing parental perceived efficacy, a dimension of family functioning
Change in Parenting Sense of Competence (PSOC) from baseline to five months | Change from baseline to five months post-intervention
  Parent report assessing parental perceived efficacy, a dimension of family functioning
Change in Parenting Sense of Competence (PSOC) from baseline to nine months | Change from baseline to nine months post-intervention
  Parent report assessing parental perceived efficacy, a dimension of family functioning
Change in Peds QL Family Impact Module from baseline to one month | Change from baseline to one month post-intervention
  Parent report assessing family functioning
Change in Peds QL Family Impact Module from baseline to five months | Change from baseline to five months post-intervention
  Parent report assessing family functioning
Change in Peds QL Family Impact Module from baseline to nine months | Change from baseline to nine months post-intervention
  Parent report assessing family functioning

CONTACTS AND LOCATIONS:
Overall Officials: Amanda R Tarullo, Ph.D., Principal Investigator — Boston University
Locations (2):
- United States (2):
  - University of Denver, Denver, Colorado
  - Boston University, Boston, Massachusetts

REFERENCES:
- [Background] Garrison MM. The feedback whirlpool of early childhood sleep and behavior problems. JAMA Pediatr. 2015 Jun;169(6):525-6. doi: 10.1001/jamapediatrics.2015.0356. No abstract available. PMID 25868054
- [Background] El-Sheikh M, Buckhalt JA, Mark Cummings E, Keller P. Sleep disruptions and emotional insecurity are pathways of risk for children. J Child Psychol Psychiatry. 2007 Jan;48(1):88-96. doi: 10.1111/j.1469-7610.2006.01604.x. PMID 17244274
- [Background] Campbell SB. Behavior problems in preschool children: a review of recent research. J Child Psychol Psychiatry. 1995 Jan;36(1):113-49. doi: 10.1111/j.1469-7610.1995.tb01657.x. PMID 7714027
- [Background] Jackson CL, Redline S, Emmons KM. Sleep as a potential fundamental contributor to disparities in cardiovascular health. Annu Rev Public Health. 2015 Mar 18;36:417-40. doi: 10.1146/annurev-publhealth-031914-122838. PMID 25785893
- [Background] LeBourgeois MK, Harsh JR. Development and psychometric evaluation of the Children's Sleep-Wake Scale<sup/> Sleep Health. 2016 Sep;2(3):198-204. doi: 10.1016/j.sleh.2016.04.001. PMID 28066802
- [Background] Shields A, Cicchetti D. Emotion regulation among school-age children: the development and validation of a new criterion Q-sort scale. Dev Psychol. 1997 Nov;33(6):906-16. doi: 10.1037//0012-1649.33.6.906. PMID 9383613
- [Background] Wilson KE, Lumeng JC, Kaciroti N, Chen SY, LeBourgeois MK, Chervin RD, Miller AL. Sleep Hygiene Practices and Bedtime Resistance in Low-Income Preschoolers: Does Temperament Matter? Behav Sleep Med. 2015;13(5):412-23. doi: 10.1080/15402002.2014.940104. Epub 2014 Sep 15. PMID 25221914
- [Background] Sivertsen B, Harvey AG, Reichborn-Kjennerud T, Torgersen L, Ystrom E, Hysing M. Later emotional and behavioral problems associated with sleep problems in toddlers: a longitudinal study. JAMA Pediatr. 2015 Jun;169(6):575-82. doi: 10.1001/jamapediatrics.2015.0187. PMID 25867179
- [Background] Shaw DS, Shelleby EC. Early-starting conduct problems: intersection of conduct problems and poverty. Annu Rev Clin Psychol. 2014;10:503-28. doi: 10.1146/annurev-clinpsy-032813-153650. PMID 24471370
- [Background] Mulraney M, Giallo R, Lycett K, Mensah F, Sciberras E. The bidirectional relationship between sleep problems and internalizing and externalizing problems in children with ADHD: a prospective cohort study. Sleep Med. 2016 Jan;17:45-51. doi: 10.1016/j.sleep.2015.09.019. Epub 2015 Oct 23. PMID 26847973